CLINICAL TRIAL: NCT01486225
Title: Exploratory Comparative Single-blind Study Evaluating Tolerability of the Silicone Bands on Medical Compression Stockings
Brief Title: Tolerance Study of the Silicone Bands on Medical Compression Stockings
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Laboratoires Innothera (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CVE401-10
Record Dates: First submitted 2011-08-10; First posted 2011-12-06 (Estimated); Last update posted 2014-08-08 (Estimated); Status verified 2012-07

CONDITIONS: Skin Lesions

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Innothera's brand Stokings (Other): Innothera's branded grip-top silicone band stokingc
  Interventions: Device: Innothera's brand Stockings
- Other than Innothera's brand (Other)
  Interventions: Other: Stockings other than Innothera's brand

INTERVENTIONS:
Device: Innothera's brand Stockings — 15 patients having used Innothera branded Stocking
  Other Names: Medical compression stockings
  Arms: Innothera's brand Stokings
Other: Stockings other than Innothera's brand — 15 patients having used any other brand than Innothera's brand stockings
  Other Names: Other Names:; Medical compression stockings
  Arms: Other than Innothera's brand

SUMMARY:
The purpose of this study is to identify the nature of skin lesions that develop on contact with the grip-top bands of medical compression stockings, which are composed mainly of silicone.

DETAILED DESCRIPTION:
To identify the nature of lesions the investigator will analyse results of the biopsys, microbiological analyses, dermatological tests.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who notified a health care professional (doctor or pharmacist) of an incident with a grip-top bands compression stocking, regardless of brand and model.
* Subjects presenting skin lesions caused by the contact with silicone-containing grip-top bands of medical compression stockings (all brands combined).
* Subjects for whom the incriminated stockings provide class 2 compression or higher.
* Subjects covered by French national health insurance.
* Subjects who give their written informed consent and who accept the constraints of the study.

Exclusion Criteria:

* Known allergy to local anesthetics (lidocaine, etc.).
* History of anaphylactic shock.
* Ongoing antihistamine treatment or having taken during the week before inclusion.
* Patient on ongoing systemic corticosteroids or having taken corticosteroids in the month before inclusion.
* Patient having used a topical corticosteroid in the area where the patch tests or prick tests will be performed during the week before inclusion.
* Phototherapy or sun exposure in the 30 days preceding the skin tests (on the back).
* Patient having concomitantly used compression stockings and a topical corticosteroid on the thighs in the 48 hours preceding lesion onset.
* List of diseases which will prevent a subject from participating in the study:
* acquired, infectious or drug-induced congenital immunosuppression (systemic corticosteroid therapy, immunosuppressives, chemotherapy),
* Congenital bullous disorder (congenital epidermolysis bullosa) or acquired bullous disorder (pemphigus, pemphigoid, dermatitis herpetiformis, linear IgA dermatosis, etc.).
* Patients with an ongoing or previous history of mental or psychiatric disorder or condition or any other factor interfering with the ability to give informed consent.
* Any major systemic disease making the conduct of the study or the interpretation of the results difficult.
* Patients with ongoing or previous history of decompensated heart failure.
* Chemotherapy or active cancer.
* Pregnancy.
* Patients participating in an ongoing clinical trial or in the exclusion period of a previous trial.
* Persons deprived of their liberty by judicial or administrative decision or persons hospitalized without their consent.
* Legally protected adults under guardianship.
* If the patient accepts the biopsy proposed in the study:
* Patient for whom a skin biopsy is contra-indicated or requiring antibiotic prophylaxis,
* Anticoagulant taken during the 24 hours before inclusion.
* Subject with history of allergy to natural or synthetic latex, chlorhexidine, known healing disorder and/or viral diseases transmissible through the blood documented by the preliminary clinical exam.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2011-11; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
nature and outcome of skin lesion caused by the silicone from the grip-top band of medical stockings | within 5 days from skin lesion started
  Patient will be followed during 5 days from the time that lessions occurs

CONTACTS AND LOCATIONS:
Overall Officials: Annick BARBAUD, MD Professor, Principal Investigator — Central Hospital, Nancy, France
Locations (1):
- Hôpitaux de Brabois CHU de Nancy, Nancy, France